CLINICAL TRIAL: NCT00936494
Title: Inferior Turbinate Reduction in Pediatric Population Failing Tonsillectomy and Adenoidectomy for Sleep Disordered Breathing (Randomized, Prospective, Controlled Study)
Brief Title: Inferior Turbinate Reduction in Pediatric Population Failing Surgery for Sleep Disordered Breathing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1137500
Record Dates: First submitted 2009-07-09; First posted 2009-07-10 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Sleep Related Breathing Disorder; Upper Airway Resistance Syndrome; Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; sleep related breathing disorder; snoring; disturbed sleeping; open mouth breathing; upper airway resistance syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring; Mouth Breathing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No inferior turbinate surgery.
- Intervention (Other): Intervention group: Cold ablation inferior turbinate reduction utilizing radiofrequency ablation surgery (CITR).
  Interventions: Procedure: Cold ablation inferior turbinate reduction

INTERVENTIONS:
Procedure: Cold ablation inferior turbinate reduction — The procedure usually takes 30 minutes and involves the surgeon inserting the coblation inferior turbinate reduction wand into the inferior turbinates and allowing for the radiofrequency cold ablation to ablate soft tissues, with a resultant thermal lesion allowing for additional soft tissue attenuation and contracture with time.
  Other Names: Radiofrequency ablation surgery; CITR
  Arms: Intervention

SUMMARY:
This study will examine whether treatment of inferior turbinates in patients with continued symptoms of obstructive sleep apnea, sleep related breathing disorder, snoring, disturbed sleeping, open mouth breathing, and upper airway resistance syndrome after tonsillectomy and adenoidectomy will improve these symptoms and should be included in the treatment paradigm for treatment of sleep related breathing disorders in infants, children, and adolescents.

DETAILED DESCRIPTION:
The question proposed by this study is one of treatment: To what extent does treatment of nasal obstruction from enlarged inferior turbinates with cold ablation inferior turbinate reduction in infants, children, and adolescents improve symptoms of obstructive sleep apnea, sleep related breathing disorder, snoring, disturbed sleeping, open mouth breathing, and upper airway resistance syndrome in patients that continue to have symptoms after tonsillectomy and adenoidectomy.

The trial seeks to provide evidence that the treatment of inferior turbinates in patients with continued symptoms of obstructive sleep apnea, sleep related breathing disorder, snoring, disturbed sleeping, open mouth breathing, and upper airway resistance syndrome after tonsillectomy and adenoidectomy will improve these symptoms and should be included in the treatment paradigm for treatment of sleep related breathing disorders in infants, children, and adolescents.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that underwent tonsillectomy and adenoidectomy for obstructive sleep apnea, sleep related breathing disorder, snoring, disturbed sleeping, open mouth breathing, and upper airway resistance syndrome with persistent symptomatology.
2. Enlarged inferior turbinates with nasal obstruction (>25%).
3. Age 0-18 years.
4. Lack of improvement of obstructive sleep apnea symptoms after maximal medical treatment with intranasal steroids in patients with symptoms of ARS and H2 blocker medication in patients with symptoms of LPR.

Exclusion Criteria:

1. Previous adenotonsillar surgery or placement of tympanostomy tubes for recurrent otitis media, tonsillitis, or sinusitis.
2. Patients with BMI > 97% for age and sex.
3. Patients with craniofacial abnormalities.
4. Patients with previous airway issues, anatomic variance from normal, mallampati class III or IV, septal deviation, choanal stenosis, and nasal stenosis.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
resolution of obstructive sleep apnea symptoms on pediatric sleep questionaire | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eliav Gov-Ari, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospitals and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No